CLINICAL TRIAL: NCT05834881
Title: Reducing Opioid and Other Drug Use in Justice-Involved Emerging Adults Using Paraprofessional Coaches (With and Without Lived Experience) to Deliver Effective Services in a Non-Treatment Setting
Brief Title: Reducing Drug Use in Justice-Involved Emerging Adults
Acronym: PEERS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chestnut Health Systems (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Tess Drazdowski, Principal Investigator, Chestnut Health Systems
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: K23DA048161 (NIH); K23DA048161 (NIH)
Record Dates: First submitted 2023-03-22; First posted 2023-04-28 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Substance-Related Disorders
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CM combined with Vocational/educational Coaching from Coaches without Lived Experience (Experimental): This group will receive contingency management (CM) combined with vocational/educational coaching from paraprofessional coaches without lived experience in community settings.
  Interventions: Behavioral: Contingency Management (CM) combined with vocational/educational coaching
- CM combined with Vocational/educational Coaching from Coaches with Lived Experience (Active Comparator): This group will receive contingency management (CM) combined with vocational/educational coaching from paraprofessional coaches with lived experience in community settings.
  Interventions: Behavioral: Contingency Management (CM) combined with vocational/educational coaching

INTERVENTIONS:
Behavioral: Contingency Management (CM) combined with vocational/educational coaching — Two evidence based practices, CM and vocational/educational coaching, will be combined and delivered by paraprofessional coaches in an intervention named PEERS (Peers Education Empowering Recovery Supports). CM uses positive reinforcement (e.g., chances to win prizes) for clients who abstain from substance use. A standardized and well-validated CM protocol will be used in the proposed study. Vocational/educational coaching assists individuals in completing educational and vocational goals. A workbook developed specifically for vocational/educational coaching in emerging adults will be used in the study.

SUMMARY:
The overarching purpose of this pilot study is to investigate an increasingly common, but under-researched, practice of employing paraprofessional coaches to improve emerging adults' access to and engagement in evidence-based substance use practices, focusing on the paraprofessional coaches' outcomes and the role of lived experience.

DETAILED DESCRIPTION:
Criminal legal system involved emerging adults are one of the highest-risk populations for opioid and other substance use and other significant problems (criminal behaviors), but they lack access to and engagement in evidence-based practices. The deleterious outcomes and long-term costs of substance use for emerging adults, communities, and society (estimated at over $740 billion annually and greater than costs for any other health problem), make this a priority. This pilot project is aimed at using paraprofessional coaches to increase engagement and access to evidence-based practices (i.e., contingency management for substance use and vocational/educational coaching) for emerging adults with substance use and criminal legal system involvement. In partnership with parole and probation, sixty emerging adults with substance use will be randomized to work with twenty paraprofessional coaches either with or without lived experience (i.e., successful substance use recovery and/or adult criminal legal system involvement). Although using peer paraprofessional coaches (those with lived experience) is becoming more popular and supported at the federal level, the outcome of this work on the paraprofessional coaches themselves, especially for emerging adults, is largely unexplored. The proposed study will use both quantitative and qualitative methods to assess feasibility and acceptability of the services and research protocols and to gain a better understanding of the impacts on both the coaches and their emerging adult clients. As substance use and poor vocational/educational attainment greatly increases the likelihood of recidivism, innovative strategies to reduce opioid and other substance use for emerging adults is critical, along with understanding the effects on the service providers (i.e., paraprofessional coaches). Aim 1: Determine the feasibility of paraprofessional coaches to deliver (with high adherence) the established interventions to emerging adults with substance use and criminal legal system involvement as part of probation and parole services, and explore differences in the delivery of the interventions based on lived experience. Aim 2: Compare emerging adult clients' engagement (attendance, completion of the intervention) and outcomes (substance use, vocational/educational attainment, criminal recidivism), when interventions are delivered by paraprofessional coaches with vs. without lived experience. Aim 3: For paraprofessional coaches delivering the interventions, examine the differences over time between those with vs. without lived experience on their own substance use symptoms and substance use relapse risk factors.

ELIGIBILITY:
There are two types of participants in this study: (1) Paraprofessional Coaches and (2) Emerging Adult Clients

Paraprofessional Coach Eligibility Criteria

Inclusion:

-Between 18-30 years old

Exclusion:

-Life threatening or unstable condition requiring treatment (e.g., suicidal/homicidal ideation)

Emerging Adult Client Eligibility Criteria

Inclusion:

* 18-26 years old
* Have current or historical lived experience with the juvenile or adult criminal legal system (e.g., probation, parole, diversion, deflection).
* Screen positive for substance use disorder

Exclusion:

* Qualifying for federal disability benefits which would preclude them from engaging in educational/vocational coaching
* Currently unhoused without a primary address
* Life threatening or unstable condition requiring treatment (e.g., suicidal/homicidal ideation)

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2023-05-26 (Actual); Primary Completion 2025-12-17 (Actual); Study Completion 2025-12-17 (Actual)

PRIMARY OUTCOMES:
Changes from baseline up to 30 months post-baseline in Paraprofessional Coach Urine Drug Screens (measured at 0, 6, 12, 18, 24, and 30 months). | Baseline to 30 months
  Number of positive drug screens from toxicology testing with paraprofessional coaches for amphetamines, barbiturates, buprenorphine, benzodiazepines, cocaine, fentanyl, methamphetamines, methylenedioxymethamphetamine (MDMA), methadone, oxycodone, phencyclidine (PCP), tetrahydrocannabinol (THC), alcohol (ETG), and morphine.
Changes from baseline to 6 months post-baseline in Emerging Adult Client Urine Drug Screens (measured at 0, 4, and 6 months). | Baseline to 6 months
  Number of positive drug screens from toxicology testing with emerging adult clients for amphetamines, barbiturates, buprenorphine, benzodiazepines, cocaine, fentanyl, methamphetamines, methylenedioxymethamphetamine (MDMA), methadone, oxycodone, phencyclidine (PCP), tetrahydrocannabinol (THC), alcohol (ETG) and morphine.

SECONDARY OUTCOMES:
Changes from baseline to 6 months post-baseline in Emerging Adult Client Abstinence Self Efficacy (measured at 0, 4, and 6 months). | Baseline to 6 months
  Levels of abstinence self-efficacy reported by emerging adult clients on the Abstinence Self Efficacy Scale.
Levels of services Emerging Adult Client Satisfaction with Treatment (measured at 4 and 6 months). | Baseline to 6 months
  Levels of satisfaction with the coaches' services reported by emerging adult clients on the Client Satisfaction Questionnaire.
Changes from baseline to 6 months post-baseline in Emerging Adult Client Vocational and Educational Attainment (measured at 0, 4, and 6 months). | Baseline to 6 months
  Advancement of vocational and educational attainment reported by emerging adult clients on the modified JCOIN Core Measures Demographics.
Changes from baseline to 6 months post-baseline in Emerging Adult Client Quality of Relationship with Paraprofessional Coach (measured at 0, 4, and 6 months). | Baseline to 6 months
  Levels of the quality of the relationship between the emerging adult client and the paraprofessional coach as reported by emerging adult clients on the Dual Role Relationship Inventory.
Changes from baseline to 6 months post-baseline in Emerging Adult Recovery Capital (measured at 0, 4, and 6 months). | Baseline to 6 months
  Levels of recovery capital as reported by emerging adult clients on the Emerging Adult Recovery Capital Scale.
Changes from baseline to 6 months post-baseline in Emerging Adult Substance Use and Problems (measured at 0, 4, and 6 months). | Baseline to 6 months
  Frequency of substance use and substance-related problems reported by emerging adult clients on the Global Appraisal of Individual Needs.
Changes from baseline to 6 months post-baseline in Emerging Adult Criminal Legal System Involvement (measured at 0, 4, and 6 months). | Baseline to 6 months
  Frequency of criminal legal system involvement reported by emerging adult clients on the Justice Community Opioid Innovation Network (JCOIN) Core Measures Justice Involvement Scale.
Changes from baseline to 6 months post-baseline in Emerging Adult Service Utilization (measured at 0, 4, and 6 months). | Baseline to 6 months
  Frequency of service utilization reported by emerging adult clients on the JCOIN Core Measures Service Utilization Scale.
Changes from client's 18th birthday to 6 months post-baseline in Emerging Adult Client Arrests. | From client's 18th birthday to 6 months post-baseline
  Number of emerging adult client arrests before and during service engagement measured via official arrest records.
Changes from client's 18th birthday to 6 months post-baseline in Emerging Adult Client Charges. | From client's 18th birthday to 6 months post-baseline
  Number of emerging adult client charges before and during service engagement measured via official arrest records.
Changes from client's 18th birthday to 6 months post-baseline in Emerging Adult Client Convictions. | From client's 18th birthday to 6 months post-baseline
  Number of emerging adult client convictions before and during service engagement measured via official arrest records.
Changes from client's 18th birthday to 6 months post-baseline in Emerging Adult Client Incarcerations. | Client's 18th birthday to 6 months
  Number of emerging adult client incarcerations before and during service engagement measured via official arrest records.
Attitudes at 6 months post-baseline in Emerging Adult Client Attitudes Toward the Services Provided (measured at 6 months). | 6 months
  Emerging adult attitudes toward the services program as measured during qualitative interviews with emerging adult clients.
Changes from baseline to 6 months in Emerging Adult Client Session Attendance and Vocational/Educational Activity Completion (measured at 1, 2, 3, 4, 5, and 6 months). | Baseline to 6 months
  Frequency of emerging adult attendance at their paraprofessional coach sessions and completion of vocational/educational coaching activities reported by paraprofessional coaches on the Session Checklist and session tape coding.
Rates of post-services Services Completion. | Post-services, an average of 6 months
  Rates of emerging adult client services completion reported by paraprofessional coaches using the Services Termination Form.
Changes from baseline to up to 30 months post-baseline in Paraprofessional Coach Abstinence Self Efficacy (measured at 0, 6, 12, 18, 24, and 30 months). | Baseline to 30 months
  Levels of abstinence self-efficacy reported by paraprofessional coaches on the Abstinence Self Efficacy Scale.
Changes from baseline to up to 30 months post-baseline in Paraprofessional Coach Attitudes Toward Medications for Opioid Use Disorder (MOUD) (measured at 0, 6, 12, 18, 24, and 30 months). | Baseline to 30 months
  Levels of attitudes toward MOUD reported by paraprofessional coaches on the JCOIN Core Measures Attitudes Toward MOUD Scale.
Changes from Baseline scores compared to up to 30 months post-baseline in Paraprofessional Coach Contingency Management (CM) Adherence (measured monthly for 30 months). | Baseline to 30 months
  Adherence to CM practices by paraprofessional coaches as measured using the CM-Therapist Adherence Measure (CM-TAM) (Self-report version and Tape Coding version).
Changes from baseline up to 30 months post-baseline in Paraprofessional Coach Client Vocational and Educational Attainment (measured at 0, 6, 12, 18, 24, and 30 months). | Baseline to 30 months
  Advancement of vocational and educational attainment reported by paraprofessional coaches on the modified JCOIN Core Measures Demographics.
Changes from baseline up to 30 months post-baseline in Paraprofessional Coach Recovery Capital (measured at 0, 6, 12, 18, 24, and 30 months). | Baseline to 30 months
  Levels of recovery capital as reported by paraprofessional coaches on the Emerging Adult Recovery Capital Scale.
Changes from baseline up to 30 months post-baseline in Paraprofessional Coach Substance Use and Problems (measured at 0, 6, 12, 18, 24, and 30 months). | Baseline to 30 months
  Frequency of substance use and substance-related problems reported by paraprofessional coaches on the Global Appraisal of Individual Needs.
Changes from baseline up to 30 months post-baseline in Paraprofessional Coach Perceptions of Acceptability of the PEERS Intervention (measured at 0, 6, 12, 18, 24, and 30 months). | Baseline to 30 months
  Levels of acceptability of the PEERS intervention, such as if participants like the intervention, as reported by paraprofessional coaches on the Acceptability of Intervention Measure (Weiner et al., 2017). Scores range from 4-20. Higher scores indicate higher levels of intervention acceptability.
Changes from baseline up to 30 months post-baseline in Paraprofessional Coach Perceptions of PEERS Intervention Appropriateness (measured at 0, 6, 12, 18, 24, and 30 months). | Baseline to 30 months
  Levels of PEERS intervention appropriateness, such as if the intervention is a good match, as reported by paraprofessional coaches on the Intervention Appropriateness Measure (Weiner et al., 2017). Scores range from 4-20. Higher scores indicate higher levels of intervention appropriateness.
Changes from baseline up to 30 months post-baseline in Paraprofessional Coach Perceptions of Feasibility of the PEERS Intervention (measured at 0, 6, 12, 18, 24, and 30 months). | Baseline to 30 months
  Levels of PEERS intervention feasibility, such as if the intervention is easy to use, as reported by paraprofessional coaches on the Feasibility of Intervention Measure (Weiner et al., 2017). Scores range from 4-20. Higher scores indicate higher levels of intervention feasibility.
Changes from baseline up to 30 months post-baseline in Paraprofessional Coach Quality of Life (measured at 0, 6, 12, 18, 24, and 30 months). | Baseline to 30 months
  Levels of quality of life reported by paraprofessional coaches on the JCOIN Core Measures Quality of Life Scale from the Patient-Reported Outcomes Measurement Information System.
Changes from post-training to post-service delivery on attitudes towards the training, supervision, and implementation of the services delivery (measured at approximately 1, 6, and 12 months). | Post-training, an average of one month, to post-service delivery of two more clients, an average of one year
  Ratings on attitudes towards the training, supervision, and implementation of the services delivery as measured by qualitative interviews with paraprofessional coaches.
Differences in themes derived from 60 audio-recorded sessions tapes varied across paraprofessional coaches, emerging adult clients, session number, and project timeline from Paraprofessional Coaches With and Without Lived Experience (measured monthly). | Across Services Delivery, an average of 6 months
  Sixty tapes from audio-recorded sessions of paraprofessional coaches with their emerging adult clients will be coded to determine themes that arise in the course of sessions to compare themes used in sessions by paraprofessional coach with and without lived experience.

CONTACTS AND LOCATIONS:
Locations (1):
- Chestnut Health Systems, Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: No